CLINICAL TRIAL: NCT03144362
Title: Unilateral and Bilateral Neurodynamic Sliding Techniques as a Means of Treating Non-compressive Sciatic Leg Pain: A Pilot Study for a Randomised Controlled Trial
Brief Title: Neurodynamic Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Purpose: Treatment
Other Study IDs: STH19135
Record Dates: First submitted 2017-05-04; First posted 2017-05-08 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Sciatic Leg Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bilateral Sliding Technique (Active Comparator)
  Interventions: Procedure: Bilateral Sliding Techniques
- Unilateral Sliding Techniques (Active Comparator)
  Interventions: Procedure: Unilateral Sliding Techniques
- Standard care (No Intervention)

INTERVENTIONS:
Procedure: Bilateral Sliding Techniques — Bilateral Sliding Techniques
  Arms: Bilateral Sliding Technique
Procedure: Unilateral Sliding Techniques — Unilateral Sliding Techniques
  Arms: Unilateral Sliding Techniques

SUMMARY:
Sciatica is a debilitating and costly condition. Prognostically, patients presenting with leg pain often have a poor recovery and some go onto have spinal surgery. However, in the absence of nerve root compression on MRI, no surgical option is viable and patients are often discharged and encouraged to self manage. Neurodynamics offers a means to treat patients with non-compressive leg pain. To date, there is no research exploring which form of neurodynamic sliding technique offers the greatest therapeutic benefit in patients presenting with sciatica. The aim of this pilot study is to calculate how many patients would be needed to run a full scale trial evaluating therapeutic efficacy. Moreover, the pilot will assess the overall workability of the study and the feasibility of patient recruitment.

DETAILED DESCRIPTION:
Patients who have given informed consent will be randomly allocated to one of three groups in a ratio of 1:1:1 (Control Group, Intervention Group 1, Intervention Group 2). Randomisation reduces selection bias and controls for unknown variables that may affect the outcome. Treatment allocation will occur through the use of sealed, opaque envelopes and will be implemented by the Graves Move More reception team as the patient attends the clinic. The reception staff will hand an opaque envelope to the subject for them to open. Randomisation undertaken by an independent third party improves internal validity. Patients will be treated according to the group they have been randomised to.

Data Collection, Analysis & Statistical Opinion Prior to undertaking the study, baseline socio-demographic data will be recorded (E.g. age, sex, weight, height, occupation and duration of symptoms). Pre and posttest outcome data will also be recorded for the Roland-Morris Disability Questionnaire (RMDQ) and Oswestry Disability Index 2.0 (ODI). Long-term data (I.e. 6-12 months post-treatment) will not be recorded as treatment effect is not being analysed as part of the pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with sciatic leg pain or dysaesthetic symptoms into one leg, below the knee who have had lumbar/sacral nerve root compression excluded through MRI
* Duration of symptoms greater than 12 weeks
* Reproduction of the patients symptoms with SLR test + passive ankle dorsiflexion
* Patients aged between 18-75 years of age (both male and female participants)

Exclusion Criteria:

* Any form of lower limb or spinal entrapment neuropathy
* Patients who have not had a lumbosacral MRI
* Any contraindications to manual therapy including; cancer, cauda equina syndrome, active inflammatory arthropathies, rapidly deteriorating neurology, spinal fracture
* Previous lumbar spinal surgery
* Inability to undertake side lying
* Patients unable to give informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Roland Morris Disability Questionnaire | 6 months
  The questionnaire will be completed prior to treatment starting and again at the conclusion of the study. Change scores will be recorded. Roland & Fairbank (2000) advise a change score of 2-3 points on the 24-item version of the RMDQ as the minimally clinically important difference (MCID).

SECONDARY OUTCOMES:
The Oxford Disability Index | 6 months
  The Oxford Disability Index (ODI) accounts for the Roland Morris Disability Questionnaire shortcomings as it is more responsive to patients presenting with more chronic, and or severe disability (Roland & Fairbank, 2000). The MCID for the ODI has been specified as 4 points (Co et al, 1993). Neither questionnaire require permission to be used in this trial Again, pre and post-test data will be recorded to calculate change scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided